CLINICAL TRIAL: NCT02878915
Title: Assessing the Interest of Ultrasound-guided Femoral Arterial Puncture for Interventional Neuro-radiology in Children
Brief Title: Ultrasound-guided Femoral Arterial Puncture for Interventional Neuro-radiology in Children
Acronym: FAP-ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RBC_2014-34
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Retrograde Femoral Catheterism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound guided femoral puncture (Active Comparator): Ultrasound guided femoral puncture
  Interventions: Device: Ultrasound guided femoral puncture
- Palpation guided femoral puncture (No Intervention): Palpation guided femoral puncture

INTERVENTIONS:
Device: Ultrasound guided femoral puncture
  Arms: Ultrasound guided femoral puncture

SUMMARY:
Using ultrasound to guide vascular catheterism in children is highly recommended for central venous access. It has been proven that central venous line is inserted faster, with fewer attempts and complications. Its interest in central arterial line insertion is less obvious. It seems to have benefits in adults, both for radial and femoral arterial insertion. But there is no study assessing the interest of ultrasound guided arterial puncture in children,.

DETAILED DESCRIPTION:
The use of ultrasound to guide vascular catheterization in children is strongly recommended for central venous vascular access by several international learned societies. In fact, studies have found a reduction in the time it takes to install the central venous line, in the number of attempts and in complications.The benefit of ultrasound to guide catheterization of the arterial network is less documented.

In children, there is an inventory of the traditional approach guided by palpation, in children in intensive care (11). The analysis of 77 femoral puncture attempts in 74 children was carried out. Arterial cannulation was successful in 73 of 77 cases (95%), but only in 60% of cases at the first attempt. Ultrasound guidance appears beneficial in adults for both arterial sites, radial and femoral. On the other hand, in children, unlike radial catheterization, there is no study evaluating the contribution of ultrasound guidance for femoral catheterization.

ELIGIBILITY:
Inclusion Criteria:

* requirement of retrograde femoral arterial catheterism

Exclusion Criteria:

* none

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Demonstrate that ultrasound guidance improves the success rate at the 1st attempt | immediate
  The success rate of catheterisation in the 1st trial will be analysed as the main criterion and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Blanc, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No